CLINICAL TRIAL: NCT03803085
Title: A Group-Based Walking Study Using WeChat to Enhance Physical Activity Among Older Adults: The Role of Social Engagement
Brief Title: A Group-Based Walking Study Using WeChat to Enhance Physical Activity Among Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brandeis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18131
Record Dates: First submitted 2018-09-24; First posted 2019-01-14 (Actual); Results first posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-10

CONDITIONS: Inactivity; Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: A total of 60 adults were recruited and randomly assigned to either the control condition (n=30) or the treatment condition (n=30). The 60 participants completed the study in one of three subgroups, with 20 participants randomly assigned to two groups (10 in the treatment group and 10 in the control group). Both conditions will use the WeChat App for use on a smartphone. The control group used the WeRun program to count their own steps. The treatment condition used the WeRun to engage in social contact and compare their steps with others in the group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Condition (Experimental): Participants only saw their own daily walking steps using the WeRun function in WeChat. They did not use WeChat to see other group members' daily steps and did not engage in social contact with their group members.
  Interventions: Behavioral: Control condition
- Treatment condition (Experimental): Participants saw their own and other group member's daily walking steps using the WeRun function in WeChat and they were able to contact the other members of their group using We Chat.
  Interventions: Behavioral: Treatment condition

INTERVENTIONS:
Behavioral: Control condition — Participants in the control group only saw their own daily walking steps using the WeChat. They did not use WeChat to see other group members' daily steps and did not contact other group members. The participants were asked to use the app every day. A message (through WeChat) was sent to remind them to use the application if they had not done so within three days.
  Arms: Control Condition
Behavioral: Treatment condition — Participants in the experimental condition used WeChat for 4 weeks to see their own and other's walking steps and also were able to contact other group members. The participants were asked to use the application every day. A message (through the group chat) was sent to remind them to use the application if they have not done so within three days.
  Arms: Treatment condition

SUMMARY:
The aim for the study is to use the function WeRun in the application WeChat to encourage physical activity and social engagement among community dwelling older adults and their family members and friends. The specific aims are to test the effectiveness of a social contact and comparison intervention for increasing regular daily physical activity among community dwelling older adults, and to examine the potential effectiveness of WeChat in cultivating social engagement and well-being among community dwelling older adults.

DETAILED DESCRIPTION:
The aim for the study is to use the function WeRun in the application WeChat to encourage physical activity and social engagement among community dwelling older adults. The investigators asked participants in the social engagement group to use the WeRun function in WeChat to track their daily walking steps and to compare their performance with their group members for 4 weeks. To encourage social engagement among their group members, the daily walking steps were calculated and the participant who has the highest step count in the group will be indicated each day.Those in the control group will only use the WeRun function in WeChat to track their own walking steps.

The investigators expected that the participants in the social contact group will walk more often and report more social activities than those in the control group, who will not compete with their peers in daily walking. To test these predictions, daily walking steps and the total walking steps per week were obtained and compared across groups. The nature and the extent of change was analyzed over the four weeks. Exercise self-efficacy was measured using a measure based on Bandura's model. Social engagement was measured using the short Lubben Social Network Scale, a self report measure of social engagement on a 12-item scale, and physical activity was measured using International Physical Activity Questionnaire (IPAQ), a self-report measure of physical activity on a 12-item scale.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are 60 or older who have a cellphone, with either android or iPhone system with data plan.
* They must be fit enough to walk for at least 20 minutes at a time.
* English speaking

Exclusion Criteria:

* Unable to walk more than 20 minutes;
* do not have smart phone with data plan.
* younger than 60

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brandeis University, Waltham, Massachusetts, United States

REFERENCES:
- [Derived] Liu Y, Lachman ME. A Group-Based Walking Study to Enhance Physical Activity Among Older Adults: The Role of Social Engagement. Res Aging. 2021 Oct-Dec;43(9-10):368-377. doi: 10.1177/0164027520963613. Epub 2020 Oct 6. PMID 33021146

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Condition: Participants saw their own and other group member's daily walking steps using the WeRun function in WeChat and they were able to contact the other members of their group using We Chat.
  Treatment condition: Participants in the treatment condition used WeChat for 4 weeks to see their own and other's walking steps and also were able to contact other group members. The participants were asked to use the application every day. A message (through the group chat) was sent to remind them to use the application if they have not done so within three days.
Period: Overall Study
Arm/Group | Control Condition | Treatment Condition
Started | 30 | 30
Completed | 28 | 28
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Treatment Condition: Participants saw their own and other group member's daily walking steps using the WeRun function in WeChat and they were able to contact the other members of their group using We Chat.
  Experimental condition: Participants in the treatment condition used WeChat for 4 weeks to see their own and other's walking steps and also were able to contact other group members. The participants were asked to use the application every day. A message (through the group chat) was sent to remind them to use the application if they have not done so within three days.
- Total: Total of all reporting groups
Arm/Group | Control Condition | Treatment Condition | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 16 | 34
  >=65 years | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (5.32) | 65.5 (5.24) | 65.4 (5.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 22 | 23 | 45
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Steps Walked
Description: Weekly average number of steps recorded with WeRun on the phone [ (averaged across 7 days at Baseline week and averaged across 7 days at Week 4 (Posttest) and averaged across 7 days at Week 8 (one month follow up)].
Time Frame: [Time Frame: Baseline (pretest) Week, Week 4 (posttest) and Week 8 (one month follow up)]
Population: Analysis population based on participants that successfully synced their WeRun and did not withdraw before the start of the study.
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Control Condition | Treatment Condition
Number analyzed (Participants) | 28 | 28
steps
  Pretest | 3992 (2388) | 4125 (2693)
  Posttest | 4171 (3122) | 5872 (3494)
  Follow-up test | 4330 (3185) | 5911 (3467)
Statistical Analysis 1: Comparison: Control Condition vs Treatment Condition; Test type: Superiority; p = 0.02, Mixed Models Analysis

2. Secondary Outcome: Social Engagement
Description: Short Lubben Social Network Scale-Revised, a self-report measure of social engagement on a 12-item scale. The total score is calculated by the sum of all the items. The total score ranges between 0 and 60, with a higher score indicating more social engagement.
Time Frame: Pretest given 1 week before the intervention and then at the posttest after the 4 week study and one month follow up
Population: Analysis population based on those who completed social engagement measurement at each testing point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Condition | Treatment Condition
Number analyzed (Participants) | 28 | 28
units on a scale
  Pretest | 35.1 (11.5) | 35.9 (11.3)
  Posttest | 37.1 (8.3) | 45.7 (11.5)
  Follow-up test | 37.7 (8.9) | 44.1 (10.8)
Statistical Analysis 1: Comparison: Control Condition vs Treatment Condition; Test type: Superiority; p = 0.03, Mixed Models Analysis

3. Secondary Outcome: Exercise Self Efficacy
Description: This scale is a self-report of exercise self-efficacy. Total score is calculated by summing the responses to each question. This scale has a range of total scores from 0-90. A higher score indicates higher self-efficacy for exercise.
Time Frame: Pretest given 1 week before the intervention and then at the posttest after the 4 week study and one month follow up
Population: Analysis population based on those who completed exercise self-efficacy measurement at each testing point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Condition | Treatment Condition
Number analyzed (Participants) | 28 | 28
units on a scale
  Pretest | 57.7 (22.8) | 60.3 (22.3)
  Posttest | 55.8 (21.8) | 67.0 (21.6)
  Follow-up test | 53.2 (21.4) | 60.3 (22.5)
Statistical Analysis 1: Comparison: Control Condition vs Treatment Condition; Test type: Superiority; p = 0.06, Mixed Models Analysis — p<0.05 was considered significant

ADVERSE EVENTS:
Time Frame: From enrollment through study completion, an average of 2 months
Description: The risks of participation were low. We included individuals whose functional health is sufficient for normal walking. We provided goals that increased their activity level, and were tailored to their current level of activity.
Arm/Group | Control Condition | Treatment Condition
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT03803085/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT03803085/ICF_001.pdf